CLINICAL TRIAL: NCT07207707
Title: A Phase 1a, Open-label, Multicenter, Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of KQB548 in Participants With Advanced Solid Malignancies With a KRAS G12D Mutation
Brief Title: A Study to Investigate the Safety and Efficacy of KQB548 in Participants With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kumquat Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQB548-101
Record Dates: First submitted 2025-09-03; First posted 2025-10-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor Malignancies
Keywords: KRAS; G12D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: KQB548

INTERVENTIONS:
Drug: KQB548 — Oral KQB548

SUMMARY:
The goal of this trial is to learn if KQB548 works to treat patients with advanced solid malignancies with a KRAS G12D mutation. It will also learn about the safety of KQB548. The main questions it aims to answer are:

* What is the safe dose of KQB548?
* Does KQB548 decrease the size of the tumor?
* What happens to KQB548 in the body?

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, locally advanced or metastatic PDAC, CRC, or NSCLC with a KRAS G12D mutation
* Progressed on, or intolerant to at least one prior line of systemic standard of care therapy
* Measurable disease according to RECIST v1.1
* Adequate organ function

Exclusion Criteria:

* Previous treatment with a KRAS G12D inhibitor or pan-RAS inhibitor
* History of intestinal disease, uncontrolled inflammatory bowel disease (e.g., Crohn's disease, Ulcerative Colitis), major esophageal or gastric surgery, or other gastrointestinal conditions (e.g., uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study intervention or result in inability to swallow oral medications
* Poorly controlled ascites and/or pleural effusion
* Requires treatment with a strong and/or moderate CYP3A inhibitor or inducer
* Requires treatment with a proton-pump inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety,Tolerability, MTD/MAD and/or RDE in the Study Population | Up to 30 months
  Safety characterized by type, incidence and severity of treatment emergent adverse events (TEAEs), SAEs, and DLTs

SECONDARY OUTCOMES:
Plasma Concentration-time curve (AUC) | Up to 30 months
Maximum plasma concentration (Cmax) | Up to 30 months
Time to maximum plasma concentration (tmax) | Up to 30 months
Overall Response Rate (ORR) | Up to 30 months
  Per RECIST v1.1
Duration of Response (DOR) | Up to 30 months
  Per RECIST v1.1
Time to Response (TTR) | Up to 30 months
  Per RECIST v1.1
Disease Control Rate (DCR) | Up to 30 months
  Per RECIST v1.1
Progression Free Survival (PFS) | Up to 30 months
  Per RECIST 1.1
Overall Survival (OS) | Up to 30 months
  Per RECIST v1.1
Peak Plasma Concentration (Cmax) in Fed and Fasted States for Food Effect | Up to 30 months
Concentration Time Curve (AUC) in Fed and Fasted States for Food Effect | Up to 30 months
Time to maximum plasma concentration (tmax) in Fed and Fasted States for Food Effect | Up to 30 months
Evaluate Changes in QTc (mSec) | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - START Midwest, Grand Rapids, Michigan
  - NEXT Oncology - Austin, Austin, Texas
  - NEXT Oncology - Dallas, Irving, Texas
  - NEXT Oncology - San Antonio, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Virginia, Fairfax, Virginia